CLINICAL TRIAL: NCT02411539
Title: A Phase I Study to Evaluate the Safety, Tolerability, and Effect of a Human Monoclonal Antibody, VRC-HIVMAB060-00-AB (VRC01), on Markers of HIV Persistence in ART-treated, HIV-infected Adults
Brief Title: Evaluating the Safety, Tolerability, and Effect of a Human Monoclonal Antibody (VRC01) on Markers of HIV Persistence in HIV-Infected Adults Receiving Antiretroviral Therapy (ART)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACTG A5342; 12003 (Registry Identifier: DAIDS-ES); UM1AI068636 (NIH)
Record Dates: First submitted 2015-04-02; First posted 2015-04-08 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2018-06

CONDITIONS: HIV Infections
Keywords: HIV; VRC01
MeSH Terms: conditions — HIV Infections | interventions — VRC01 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: VRC01 followed by placebo (Experimental): Participants received an infusion of VRC01 at Day 0 and Week 3 and an infusion of placebo (normal saline) at Weeks 6 and 9.
  Interventions: Biological: VRC01; Biological: Placebo
- Arm B: placebo followed by VRC01 (Experimental): Participants received an infusion of placebo (normal saline) at Day 0 and Week 3 and an infusion of VRC01 at Weeks 6 and 9.
  Interventions: Biological: VRC01; Biological: Placebo

INTERVENTIONS:
Biological: VRC01 — 40 mg/kg of VRC01 administered as an intravenous infusion over about 30 to 60 minutes using a volumetric pump
  Other Names: VRC-HIVMAB060-00-AB
Biological: Placebo — Normal saline administered as an intravenous infusion over about 30 to 60 minutes using a volumetric pump

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability, and effect of an experimental human monoclonal antibody (mAb), VRC-HIVMAB060-00-AB (VRC01), in adults infected with HIV who were receiving antiretroviral therapy (ART).

DETAILED DESCRIPTION:
Monoclonal antibodies (mAbs) have been developed as treatment for a variety of conditions including cancer, autoimmune disorders, and infections. mAbs may also be a potential treatment for people infected with HIV. The purpose of this study was to evaluate the safety and tolerability of an experimental human mAb, VRC-HIVMAB060-00-AB (VRC01), in HIV-infected adults receiving ART. Study researchers will also evaluate the effect of VRC01 on the number of infected cells containing unspliced HIV-1 transcripts in the blood in participants.

This study enrolled HIV-infected people 18 to 65 years old, who had been receiving ART for at least 2 years and who had a CD4+ count of 200 cells/mm^3 or greater. Participants were randomly assigned to Arm A or Arm B. Participants in Arm A received an intravenous (IV) infusion of VRC01 at Day 0 and Week 3 and an IV infusion of placebo (normal saline) at Weeks 6 and 9. Participants in Arm B received an IV infusion of placebo (normal saline) at Day 0 and Week 3 and an IV infusion of VRC01 at Weeks 6 and 9. Participants recorded their temperature and symptoms for 3 days after each infusion. Study visits occured at study entry (Day 0), and Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 15, 18, and 30. Study visits included physical examinations, clinical assessments, and blood collection.

The primary safety outcome for this study was descriptive and assessed the occurrence of Grade ≥ 3 AEs including signs/symptoms, lab toxicities, and/or clinical events that are possibly, probably, or definitely related to study treatment (as judged by the core team, blinded to treatment arm) at any time from the initial dose of study treatment to the end of study follow-up. Since this outcome is descriptive, no statistical significance testing was performed.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any FDA-approved rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV or E/CIA tests, or by HIV-1 antigen, or plasma HIV-1 RNA assay. More information on this criterion is available in the protocol.
* Received continuous ART for at least 2 years (defined as no interruptions longer than 14 consecutive days) and with no changes in the components of the ART for at least 90 days prior to study entry
* CD4+ cell count greater than or equal to 200 cells/mm^3 obtained within 60 days prior to study entry in a clinical laboratory improvement amendments (CLIA)-certified laboratory
* Plasma HIV-1 RNA below the limit of detection of the FDA-approved assays (limit of detection: 75, 50, 40 or 20 copies/mL) for greater than or equal to 2 years on ART. Participants must have had at least one documented HIV-1 RNA less than the limit of detection 12-24 months prior to study entry and at least one HIV-1 RNA less than the limit of detection within 12 months prior to study entry. All available HIV-1 RNA measurements must have been below the assay limit of detection during the 2 years prior to study entry except as allowed by the following note. NOTE: A single unconfirmed plasma HIV-1 RNA greater than the limit of detection but less than 200 copies/mL within 6-24 months was allowed if followed by a subsequent value below the limit of detection.
* Plasma HIV-1 RNA level of less than 40 copies/mL obtained by the Abbott Real-time HIV assay (m2000) or less than 20 copies/mL obtained by the Roche COBAS Taqman HIV-1 v2.0 assay within 60 days prior to entry
* The following laboratory values obtained within 60 days prior to entry by any U.S. laboratory that has a CLIA certification or its equivalent.

  * Absolute neutrophil count (ANC) greater than or equal to 750 cells/mm^3
  * Hemoglobin greater than or equal to 11.0 g/dL for men and greater than or equal to 10.0 g/dL for women
  * Platelet count greater than or equal to 100,000/mm^3
  * Creatinine clearance greater than or equal to 60 mL/min estimated by the Cockcroft-Gault equation. NOTE: A program for calculating creatinine clearance by the Cockcroft-Gault method is available on www.fstrf.org.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) (SGPT) less than or equal to 2.0 times upper limit of normal (ULN)
* Hepatitis C virus (HCV) antibody negative result within 60 days prior to study entry or, if the HCV antibody result is positive, a negative HCV RNA result within 60 days prior to study entry
* Negative HBsAg result obtained within 60 days prior to study entry
* Ability and willingness of participant to provide informed consent
* Females of reproductive potential (women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy, or bilateral oophorectomy and/or bilateral salpingectomy), needed a negative serum or urine pregnancy test within 48 hours prior to study entry. NOTE: Acceptable documentation of hysterectomy and bilateral oophorectomy, bilateral salpingectomy, tubal micro-inserts, partner who has undergone vasectomy, and menopause is participant-reported history.
* All participants must have agreed not to participate in the conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the participant/partner must use at least one reliable form of contraception (condoms, with or without a spermicidal agent; a diaphragm or cervical cap with spermicide; an intrauterine device (IUD); or hormone-based contraceptive), while receiving study treatment and for 12 weeks after stopping study treatment
* Documentation of the availability of the following stored samples from the screening visit: peripheral blood mononuclear cell (PBMC) for CD4+ T-cell associated HIV-1 RNA, DNA assay and plasma for HIV-1 SCA. Sites must receive confirmation from the processing lab via phone, email, or fax, that specimens have been entered into the AIDS Clinical Trials Group (ACTG) Laboratory Data Management System (LDMS).

Exclusion Criteria:

* Previous receipt of humanized or human monoclonal antibody (licensed or investigational)
* Weight greater than 115 kg or less than 53 kg
* Acute or ongoing AIDS-defining illness within 60 days prior to study entry
* History of a severe allergic reaction with generalized urticarial, angioedema, or anaphylaxis within 2 years of study entry
* Currently breastfeeding or pregnant
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Acute or serious illness that, in the opinion of the site investigator, requires systemic treatment and/or hospitalization within 60 days prior to entry
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 60 days prior to study entry. NOTE: Participants receiving stable physiologic doses of glucocorticoids, defined as the equivalent of prednisone less than or equal to 10 mg/day, will not be excluded. Stable physiologic glucocorticoid doses should not be discontinued for the duration of the study. In addition, participants receiving inhaled or topical corticosteroids will not be excluded.
* Treatment for hepatitis C within 24 weeks of study entry
* Vaccinations within 7 days prior to the screening, pre-entry, or study entry visits. NOTE: Participants are encouraged to get routine vaccinations, such as seasonal influenza vaccine more than 7 days prior to screening or between screening and pre-entry visits (outside of the 7-day window above).
* Initiation of ART during acute HIV-1 infection (as determined by the site investigator by history and/or available medical records)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Riddler, MD, MPH, Study Chair — Pitt CRS
Locations (13):
- United States (13):
  - UCSD Antiviral Research Center CRS, San Diego, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Ohio State University CRS, Columbus, Ohio
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Houston AIDS Research Team CRS, Houston, Texas
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Derived] Riddler SA, Zheng L, Durand CM, Ritz J, Koup RA, Ledgerwood J, Bailer RT, Koletar SL, Eron JJ, Keefer MC, Macatangay BJC, Cyktor JC, Mellors JW; AIDS Clinical Trials Group A5342 Protocol Team. Randomized Clinical Trial to Assess the Impact of the Broadly Neutralizing HIV-1 Monoclonal Antibody VRC01 on HIV-1 Persistence in Individuals on Effective ART. Open Forum Infect Dis. 2018 Oct 20;5(10):ofy242. doi: 10.1093/ofid/ofy242. eCollection 2018 Oct. PMID 30364428
- See also: To grade diagnoses, signs and symptoms, and laboratory results, sites referred to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.0, November 2014 — http://rsc.tech-res.com/safetyandpharmacovigilance/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant enrolled to the study on August 25th, 2015 and the last participant enrolled on March 4th, 2016. A total of 13 U.S. sites enrolled participants.
Groups:
- Arm A: VRC01 Followed by Placebo: Participants received an infusion of VRC01 at Day 0 and Week 3 and an infusion of placebo at Weeks 6 and 9.
  VRC01: 40 mg/kg of VRC01 administered as an intravenous infusion over about 30 to 60 minutes using a volumetric pump
  Placebo: Normal saline administered as an intravenous infusion over about 30 to 60 minutes using a volumetric pump
- Arm B: Placebo Followed by VRC01: Participants received an infusion of placebo at Day 0 and Week 3 and an infusion of VRC01 at Weeks 6 and 9.
  VRC01: 40 mg/kg of VRC01 administered as an intravenous infusion over about 30 to 60 minutes using a volumetric pump
  Placebo: Normal saline administered as an intravenous infusion over about 30 to 60 minutes using a volumetric pump
Period: Overall Study
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Confounding medical condition | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01 | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12) | 52 (11) | 48 (12)
Age, Customized [Count of Participants; unit: Participants] — Age at enrollment, categorized
  Participants
    18-29 years | 3 | 2 | 5
    30-39 years | 4 | 1 | 5
    40-49 years | 4 | 2 | 6
    50+ years | 9 | 15 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 17 | 20 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-hispanic | 13 | 14 | 27
  Black non-hispanic | 3 | 4 | 7
  Hispanic (regardless of race) | 4 | 2 | 6
IV drug history, categorical [Count of Participants; unit: Participants]
  Never | 19 | 18 | 37
  Previously | 1 | 2 | 3
BMI, categorical [Count of Participants; unit: Participants] — Categories from entry visit
  Participants
    Underweight (<18 kg/m^2) | 1 | 0 | 1
    Normal (18 - <25 kg/m^2) | 4 | 11 | 15
    Overweight (25 - <30 kg/m^2) | 10 | 6 | 16
    Obese (30+ kg/m^2) | 5 | 3 | 8
Plasma HIV-1 RNA, categorical [Count of Participants; unit: Participants] — Categorization of the result from the entry visit
  Participants
    < 40 copies/mL | 20 | 20 | 40
    >= 40 copies/mL | 0 | 0 | 0
CD4+ T-Cell Count, categorical [Count of Participants; unit: Participants] — Categorization of the average results from the screening and entry visits
  Participants
    200 - <350 cells/mm^3 | 0 | 2 | 2
    350 - <500 cells/mm^3 | 3 | 2 | 5
    >= 500 cells/mm^3 | 17 | 16 | 33
Creatinine clearance, categorical [Count of Participants; unit: Participants] — Categorization of the average results from the screening and entry visits
  Participants
    50 - 90 mL/min | 4 | 9 | 13
    > 90 mL/min | 16 | 11 | 27
Cell-associated HIV-1 RNA/DNA Ratio [Median (Inter-Quartile Range); unit: log10 ratio] — Population: Geometric average of screening and entry results. Results were not available for two participants
  log10 ratio
    number analyzed (Participants) | 19 | 19 | 38
    (all) | -1.35 [-1.63 to -1.02] | -1.51 [-1.69 to -1.30] | -1.45 [-1.63 to -1.17]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Grade 3 or Greater, Treatment Related, Adverse Event (AE)
Description: Refer to detailed description in the protocol section.
  Includes signs/symptoms, lab toxicities, and/or clinical events that are possibly, probably, or definitely related to study treatment (as judged by the core team, blinded to treatment arm) at any time from the initial dose of VRC01 to end of study follow-up. This analysis was primarily descriptive and no significance testing was performed.
Time Frame: Measured from study treatment initiation to study discontinuation (study duration is 30 weeks)
Population: Includes all available follow-up for all participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

2. Primary Outcome: Change in Cell-associated HIV-1 RNA/DNA Ratio in Total CD4+ Cells
Description: Change from baseline (geometric average of screening and entry results) to week 6 in log10 transformed cell-associated HIV-1 RNA/DNA ratio in total CD4+ cells
Time Frame: Screening, entry and week 6
Population: Analysis of participants with available results for the change in cell-associated HIV-1 RNA/DNA ratio in total CD4+ cells. All participants received at least one dose of the randomized treatment assigned. No participants received the incorrect treatment.
Measure: Median (Inter-Quartile Range); unit: log10 ratio
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 18 | 19
log10 ratio | 0.05 [-0.03 to 0.33] | -0.08 [-0.24 to 0.37]
Statistical Analysis 1: Comparison: Arm A: VRC01 Followed by Placebo vs Arm B: Placebo Followed by VRC01; The primary efficacy analysis compared the change in cell-associated HIV-1 RNA/DNA ratio (log-transformed) from baseline to week 6 between the two randomized arms, testing the null hypothesis of no difference in changes in cell-associated HIV-1 RNA/DNA ratio between the two arms using a Wilcoxon rank sum test at 10% significance level; Test type: Superiority — Assuming that a common standard deviation of change (measured as difference of log10 transformed HIV-1 RNA/DNA ratios) in both arms was 0.30, with a sample size of 36 evaluable participants (18 in each arm), the study had 88% power to detect an effect size of 0.30 log10 (2-fold) in change of cell-associated HIV-1 RNA/DNA from baseline to week 6 using a two-sided Wilcoxon rank sum test at 10% type I error rate assuming a normal distribution; p = 0.16, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon rank sum test at 10% significance level. Not adjusted for multiple comparisons

3. Secondary Outcome: Number of Participants With Premature Treatment Discontinuation, for Reasons Related to Study Treatment
Description: Study treatment was taken from entry through week 12 - this outcome assesses the number of participants who permanently and prematurely discontinued study treatment due to reasons related to the study treatment
Time Frame: Measured from study treatment initiation to study treatment discontinuation (study treatment dispensed through week 12)
Population: All participants who received at least one infusion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

4. Secondary Outcome: Change in Cell-associated HIV-1 RNA/DNA Ratio in Total CD4+ Cells - Last Value Carried Forward (LVCF)
Description: Change from baseline (geometric average of screening and entry results) to week 6 in cell-associated HIV-1 RNA/DNA ratio in total CD4+ cells, using a last value carried forward approach if week 6 cell-associated HIV-1 RNA/DNA ratio was missing. In the event that the week 6 value was missing, the week 3 value was carried forward to be used. This comparison is the change from the average of screening and entry results to the week 6 value (if available), and if week 6 result was not available, the week 3 value was used instead of the week 6 value.
Time Frame: Screening, entry, week 3 and week 6 (week 3 used as LVCF if necessary)
Population: Analysis of participants with available results for the change in cell-associated HIV-1 RNA/DNA ratio in total CD4+ cells, carrying last available result forward if missing at week 6
Measure: Median (Inter-Quartile Range); unit: log10 ratio
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 19 | 19
log10 ratio | 0.06 [-0.03 to 0.53] | -0.08 [-0.24 to 0.37]

5. Secondary Outcome: Change in Cell-associated HIV-1 RNA/DNA Ratio in Total CD4+ Cells - Across Arms
Description: Summary of within-participant change across treatment arms from the pre-VRC01 time point to the post-VRC01 time point. For Arm A, the pre-VRC01 time point used was the baseline measure (geometric average of screening and entry results) and the post-VRC01 time point was the week 6 measure. For Arm B, the pre-VRC01 time point used was the week 6 measure and the post-VRC01 time point was the week 12 measure. Change in CA-RNA/DNA ratio was calculated on the log10 scale.
Time Frame: Screening, entry and weeks 6 and 12
Population: Analysis of all participants with available pre- and post-VRC01 cell-associated RNA/DNA ratio results available. Participants from Arm A must have had results at entry and week 6. Participants from Arm B must have had results from week 6 and week 12.
Measure: Median (Inter-Quartile Range); unit: log10 ratio
Groups:
- Across Arms: Compare the pre-VRC01 and post-VRC01 time points across randomized Arms A/B. Arm A participants received an infusion of VRC01 at Day 0 and Week 3 and an infusion of placebo at Weeks 6 and 9. Arm B participants received an infusion of placebo at Day 0 and Week 3 and an infusion of VRC01 at Weeks 6 and 9. This group is to identify analyses that were assessed across randomized arms between the pre- and post-VRC01 time points.
Arm/Group | Across Arms
Number analyzed (Participants) | 37
log10 ratio | 0.09 [-0.22 to 0.33]

6. Secondary Outcome: Cell-associated HIV-1 RNA in Total CD4+ Cells
Description: Testing priority was given to samples from screening, entry and weeks 3, 6, 9 and 12. Baseline values are the geometric mean of screening and entry results. Testing of specimens at weeks 1, 4, 7, 10, 15, 18 and 30 has not been performed. The study team has decided in favor of saving these samples for future research purposes.
Time Frame: Measured at screening, entry, weeks 1, 3, 4, 6, 7, 9, 10, 12, 15, 18 and 30
Population: Analysis of participants with available cell-associated HIV-1 RNA results
Measure: Median (Inter-Quartile Range); unit: log10 copies/million CD4
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
log10 copies/million CD4
  Baseline: number analyzed (Participants) | 19 | 19
  Baseline | 1.60 [0.90 to 2.09] | 1.38 [0.90 to 2.03]
  Week 3: number analyzed (Participants) | 19 | 19
  Week 3 | 1.62 [0.87 to 2.09] | 1.56 [0.71 to 1.82]
  Week 6: number analyzed (Participants) | 18 | 19
  Week 6 | 1.48 [1.11 to 2.10] | 1.41 [0.99 to 1.90]
  Week 9: number analyzed (Participants) | 18 | 19
  Week 9 | 1.56 [1.14 to 1.90] | 1.56 [0.74 to 1.89]
  Week 12: number analyzed (Participants) | 18 | 19
  Week 12 | 1.62 [0.73 to 2.03] | 1.51 [0.76 to 2.10]

7. Secondary Outcome: Cell-associated HIV-1 DNA in Total CD4+ Cells
Description: as for outcome 6
Time Frame: Measured at screening, entry, weeks 1, 3, 4, 6, 7, 9, 10, 12, 15, 18 and 30
Population: Analysis of participants with available cell-associated HIV-1 DNA results
Measure: Median (Inter-Quartile Range); unit: log10 copies/million CD4
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
log10 copies/million CD4
  Baseline: number analyzed (Participants) | 20 | 19
  Baseline | 3.05 [2.42 to 3.20] | 3.00 [2.53 to 3.18]
  Week 3: number analyzed (Participants) | 20 | 19
  Week 3 | 2.99 [2.50 to 3.15] | 2.89 [2.61 to 3.00]
  Week 6: number analyzed (Participants) | 19 | 19
  Week 6 | 2.99 [2.46 to 3.07] | 2.92 [2.54 to 3.07]
  Week 9: number analyzed (Participants) | 19 | 19
  Week 9 | 2.96 [2.46 to 3.23] | 2.91 [2.57 to 3.15]
  Week 12: number analyzed (Participants) | 19 | 19
  Week 12 | 3.01 [2.70 to 3.17] | 2.90 [2.55 to 3.12]

8. Secondary Outcome: Cell-associated HIV-1 RNA/DNA Ratio in Total CD4+ Cells
Description: as for outcome 6
Time Frame: Measured at screening, entry, weeks 1, 3, 4, 6, 7, 9, 10, 12, 15, 18 and 30
Population: Analysis of participants with available cell-associated HIV-1 RNA/DNA ratio
Measure: Median (Inter-Quartile Range); unit: log10 ratio
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
log10 ratio
  Baseline: number analyzed (Participants) | 19 | 19
  Baseline | -1.35 [-1.63 to -1.02] | -1.51 [-1.69 to -1.30]
  Week 3: number analyzed (Participants) | 19 | 19
  Week 3 | -1.29 [-1.84 to -0.74] | -1.38 [-1.57 to -1.11]
  Week 6: number analyzed (Participants) | 18 | 19
  Week 6 | -1.28 [-1.54 to -0.88] | -1.44 [-1.78 to -1.19]
  Week 9: number analyzed (Participants) | 18 | 19
  Week 9 | -1.37 [-1.55 to -1.06] | -1.40 [-1.80 to -1.02]
  Week 12: number analyzed (Participants) | 18 | 19
  Week 12 | -1.42 [-1.80 to -1.04] | -1.33 [-1.87 to -1.09]

9. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA by Single Copy Assay (SCA) Below Assay Lower Limit
Description: The analysis of HIV-1 RNA SCA assessed the number of participants below the assay lower limit (1 copy/mL) at each measurement week. Specific specimens and time points were targeted based on Arm. Samples were not tested for Arm A at the Week 7 and Week 10 time points. Samples were not tested for Arm B at the Week 1 and Week 4 time points.
  Testing of specimens at weeks 15, 18 and 30 has not been performed. The study team has decided in favor of saving these samples for future research purposes.
Time Frame: Measured at screening, entry and weeks 1, 3, 4, 6, 7, 9, 10, 12, 15, 18 and 30
Population: Analysis of participants with available SCA results
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
Participants
  Screening | 13 | 12
  Entry | 8 | 10
  Week 1: number analyzed (Participants) | 20 | 0
  Week 1 | 9 |
  Week 3 | 9 | 11
  Week 4: number analyzed (Participants) | 19 | 0
  Week 4 | 11 |
  Week 6: number analyzed (Participants) | 19 | 19
  Week 6 | 11 | 12
  Week 7: number analyzed (Participants) | 0 | 19
  Week 7 |  | 11
  Week 9: number analyzed (Participants) | 18 | 19
  Week 9 | 13 | 9
  Week 10: number analyzed (Participants) | 0 | 19
  Week 10 |  | 11
  Week 12: number analyzed (Participants) | 19 | 19
  Week 12 | 11 | 13

10. Secondary Outcome: CD4+ T-cell Counts
Description: Baseline measure represents the average of screening and entry results
Time Frame: Measured at screening, entry and weeks 6, 12, 18 and 30
Population: Analysis of all participants with available CD4+ results
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
cells/mm^3
  Baseline | 701 [594 to 952] | 685 [535 to 843]
  Week 6: number analyzed (Participants) | 19 | 19
  Week 6 | 709 [564 to 995] | 697 [532 to 807]
  Week 12: number analyzed (Participants) | 19 | 18
  Week 12 | 734 [616 to 886] | 671 [513 to 873]
  Week 18: number analyzed (Participants) | 19 | 19
  Week 18 | 709 [529 to 885] | 672 [475 to 844]
  Week 30: number analyzed (Participants) | 18 | 19
  Week 30 | 750 [612 to 1025] | 712 [486 to 806]

11. Secondary Outcome: CD8+ T-cell Counts
Description: Baseline measure represents the average of screening and entry results
Time Frame: Measured at screening, entry and weeks 6, 12, 18 and 30
Population: Analysis of all participants with available CD8+ results
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
cells/mm^3
  Baseline | 801 [490 to 1210] | 617 [480 to 744]
  Week 6: number analyzed (Participants) | 19 | 19
  Week 6 | 688 [469 to 977] | 614 [481 to 825]
  Week 12: number analyzed (Participants) | 19 | 18
  Week 12 | 649 [508 to 1039] | 620 [439 to 852]
  Week 18: number analyzed (Participants) | 19 | 19
  Week 18 | 766 [495 to 1214] | 665 [421 to 766]
  Week 30: number analyzed (Participants) | 18 | 19
  Week 30 | 731 [551 to 990] | 655 [436 to 740]

12. Secondary Outcome: Total/Inducible Virus Recovery - Stimulated HIV-1 RNA
Description: As part of the total virus recovery assay, results for stimulated HIV-1 RNA (copies/mL) are generated
Time Frame: Measured at pre-entry, week 6 and week 12
Population: Includes all participants with available stimulated HIV-1 RNA results from virus recovery assay
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 19 | 19
log10 copies/mL
  Pre-entry | 2.83 [1.81 to 3.16] | 2.85 [2.28 to 3.49]
  Week 6 | 2.74 [2.31 to 3.41] | 3.12 [2.11 to 3.54]
  Week 12 | 2.74 [2.53 to 3.18] | 2.63 [2.27 to 3.47]

13. Secondary Outcome: Total/Inducible Virus Recovery - Unstimulated HIV-1 RNA
Description: As part of the total virus recovery assay, results for unstimulated HIV-1 RNA (copies/mL) are generated
Time Frame: Measured at pre-entry, week 6 and week 12
Population: Includes all participants with available unstimulated HIV-1 RNA results from virus recovery assay
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
log10 copies/mL
  Pre-entry: number analyzed (Participants) | 19 | 19
  Pre-entry | 1.00 [0.50 to 1.86] | 1.00 [0.00 to 1.81]
  Week 6: number analyzed (Participants) | 19 | 19
  Week 6 | 1.44 [0.71 to 1.95] | 0.92 [0.00 to 1.61]
  Week 12: number analyzed (Participants) | 18 | 19
  Week 12 | 1.25 [0.50 to 1.90] | 1.53 [1.00 to 2.01]

14. Secondary Outcome: Total/Inducible Virus Recovery - Stimulated to Unstimulated HIV-1 RNA Ratio
Description: As part of the total virus recovery assay, results for stimulated and unstimulated HIV-1 RNA (copies/mL) are generated. At each time point, the ratio of the stimulated to unstimulated HIV-1 RNA was calculated.
Time Frame: Measured at pre-entry, week 6 and week 12
Population: Includes all participants with available stimulated/unstimulated HIV-1 RNA results from virus recovery assay
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
ratio
  Pre-entry: number analyzed (Participants) | 19 | 19
  Pre-entry | 16.73 [4.76 to 104.29] | 25.49 [8.12 to 115.48]
  Week 6: number analyzed (Participants) | 19 | 19
  Week 6 | 21.03 [5.58 to 78.37] | 40.50 [10.77 to 759.42]
  Week 12: number analyzed (Participants) | 18 | 19
  Week 12 | 34.12 [5.57 to 93.90] | 16.09 [9.00 to 43.11]

15. Secondary Outcome: Total/Inducible Virus Recovery - Stimulated Cell Fluor
Description: As part of the total virus recovery assay, results for stimulated cell fluor (light units) are generated.
Time Frame: Measured at pre-entry, week 6 and week 12
Population: Includes all participants with available stimulated cell fluor results from virus recovery assay
Measure: Median (Inter-Quartile Range); unit: million light units
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 19 | 19
million light units
  Pre-entry | 25.86 [22.14 to 30.42] | 26.05 [21.42 to 30.09]
  Week 6 | 24.68 [22.00 to 30.09] | 26.13 [21.79 to 29.81]
  Week 12 | 27.38 [22.12 to 31.25] | 26.97 [22.57 to 32.01]

16. Secondary Outcome: Total/Inducible Virus Recovery - Unstimulated Cell Fluor
Description: As part of the total virus recovery assay, results for unstimulated cell fluor (light units) are generated.
Time Frame: Measured at pre-entry, week 6 and week 12
Population: Includes all participants with available unstimulated cell fluor results from virus recovery assay
Measure: Median (Inter-Quartile Range); unit: million light units
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
million light units
  Pre-entry: number analyzed (Participants) | 19 | 19
  Pre-entry | 6.86 [5.70 to 13.34] | 5.87 [4.57 to 6.93]
  Week 6: number analyzed (Participants) | 19 | 19
  Week 6 | 6.39 [4.94 to 8.01] | 6.22 [5.00 to 8.76]
  Week 12: number analyzed (Participants) | 18 | 19
  Week 12 | 8.53 [6.20 to 12.16] | 6.27 [5.05 to 8.38]

17. Secondary Outcome: Total/Inducible Virus Recovery - Stimulated to Unstimulated Cell Fluor Ratio
Description: As part of the total virus recovery assay, results for stimulated and unstimulated cell fluor (light units) are generated. At each time point, the ratio of the stimulated to unstimulated cell fluor was calculated.
Time Frame: Measured at pre-entry, week 6 and week 12
Population: Includes all participants with available stimulated/unstimulated cell fluor results from virus recovery assay
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
ratio
  Pre-entry: number analyzed (Participants) | 19 | 19
  Pre-entry | 2.91 [2.14 to 4.65] | 4.32 [3.60 to 5.13]
  Week 6: number analyzed (Participants) | 19 | 19
  Week 6 | 4.20 [3.04 to 4.78] | 3.87 [3.36 to 5.49]
  Week 12: number analyzed (Participants) | 18 | 19
  Week 12 | 3.33 [2.16 to 4.62] | 3.76 [3.52 to 4.38]

18. Secondary Outcome: Total/Inducible Virus Recovery - Percentage of Total CD4 Yield
Description: As part of the total virus recovery assay, results for %tCD4 yield are generated.
Time Frame: Measured at pre-entry, week 6 and week 12
Population: Includes all participants with available %tCD4 yield results from virus recovery assay
Measure: Median (Inter-Quartile Range); unit: percentage of Total CD4 Yield
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 19 | 19
percentage of Total CD4 Yield
  Pre-entry | 25.35 [20.00 to 32.17] | 22.00 [19.00 to 27.00]
  Week 6 | 25.00 [18.00 to 32.14] | 22.38 [17.65 to 33.33]
  Week 12 | 25.00 [21.00 to 30.32] | 22.58 [18.81 to 29.00]

19. Secondary Outcome: Change in Total/Inducible Virus Recovery - Stimulated HIV-1 RNA
Description: As part of the total virus recovery assay, results for stimulated HIV-1 RNA (copies/mL) are generated. The change from the pre-treatment time point to week 6 was assessed as a fold change (week 6 / pre-entry)
Time Frame: Measured at pre-entry, week 6
Population: Includes all participants with available stimulated HIV-1 RNA results from virus recovery assay at pre-entry and week 6 time points
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 19 | 19
fold change | 0.74 [0.31 to 8.38] | 1.32 [0.30 to 1.99]

20. Secondary Outcome: Change in Total/Inducible Virus Recovery - Unstimulated HIV-1 RNA
Description: As part of the total virus recovery assay, results for unstimulated HIV-1 RNA (copies/mL) are generated. The change from the pre-treatment time point to week 6 was assessed as a fold change (week 6 / pre-entry)
Time Frame: Measured at pre-entry, week 6
Population: Includes all participants with available unstimulated HIV-1 RNA results from virus recovery assay at pre-entry and week 6 time points
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 19 | 19
fold change | 1.37 [1.00 to 2.11] | 1.00 [0.19 to 2.42]

21. Secondary Outcome: Change in Total/Inducible Virus Recovery - Stimulated to Unstimulated HIV-1 RNA Ratio
Description: As part of the total virus recovery assay, results for stimulated and unstimulated HIV-1 RNA (copies/mL) are generated. At each time point, the ratio of the stimulated to unstimulated HIV-1 RNA was calculated. The fold change of this ratio from pre-entry to the week 6 time point was calculated for each arm (week 6 / pre-entry)
Time Frame: Measured at pre-entry and week 6
Population: Includes all participants with available stimulated/unstimulated HIV-1 RNA results from virus recovery assay
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 19 | 19
fold change | 0.69 [0.20 to 3.71] | 0.85 [0.21 to 12.38]

22. Secondary Outcome: Change in Total/Inducible Virus Recovery - Stimulated Cell Fluor
Description: As part of the total virus recovery assay, results for stimulated cell fluor (light units) are generated. The fold change from pre-entry to the week 6 time point was calculated for each arm (week 6 / pre-entry)
Time Frame: Measured at pre-entry, week 6
Population: Includes all participants with available stimulated cell fluor results from virus recovery assay at pre-entry and week 6 time points
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 19 | 19
fold change | 0.97 [0.91 to 1.09] | 0.97 [0.92 to 1.05]

23. Secondary Outcome: Change in Total/Inducible Virus Recovery - Unstimulated Cell Fluor
Description: As part of the total virus recovery assay, results for unstimulated cell fluor (light units) are generated. The fold change from pre-entry to the week 6 time point was calculated for each arm (week 6 / pre-entry)
Time Frame: Measured at pre-entry, week 6
Population: Includes all participants with available unstimulated cell fluor results from virus recovery assay at pre-entry and week 6 time points
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 19 | 19
fold change | 0.93 [0.66 to 1.15] | 1.12 [1.02 to 1.39]

24. Secondary Outcome: Change in Total/Inducible Virus Recovery - Stimulated to Unstimulated Cell Fluor Ratio
Description: As part of the total virus recovery assay, results for stimulated and unstimulated cell fluor (light units) are generated. At each time point, the ratio of the stimulated to unstimulated cell fluor was calculated. The fold change of this ratio from pre-entry to the week 6 time point was calculated for each arm (week 6 / pre-entry)
Time Frame: Measured at pre-entry, week 6
Population: Includes all participants with available stimulated/unstimulated cell fluor results from virus recovery assay at pre-entry and week 6 time points
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 19 | 19
fold change | 1.08 [0.84 to 1.64] | 0.85 [0.73 to 1.08]

25. Secondary Outcome: Change in Total/Inducible Virus Recovery - Percentage of Total CD4 Yield
Description: As part of the total virus recovery assay, results for %tCD4 yield are generated. The fold change from pre-entry to the week 6 time point was calculated for each arm (week 6 / pre-entry)
Time Frame: Measured at pre-entry, week 6
Population: Includes all participants with available %tCD4 yield results from virus recovery assay at pre-entry and week 6 time points
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 19 | 19
fold change | 1.00 [0.81 to 1.41] | 1.06 [0.77 to 1.27]

26. Secondary Outcome: VRC01 Antibody Level
Description: Summarize the pharmacokinetics (PK) of two infusions of VRC01 during study follow up
  Specific specimens and time points were targeted for testing based on Arm. Samples for Arm A were not tested for the Week 6 and Week 9 post-infusion time points. Samples for Arm B were not tested for the Week 0 and Week 3 post-infusion time points.
Time Frame: Measured at entry and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 15, 18 and 30
Population: Analysis of all participants with available results.
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
ug/mL
  Week 0 - Pre-Infusion | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]
  Week 0 - Post-Infusion: number analyzed (Participants) | 20 | 0
  Week 0 - Post-Infusion | 1726.2 [1492.5 to 1950.3] |
  Week 1 | 259.9 [213.0 to 297.5] | 0.1 [0.1 to 0.1]
  Week 2: number analyzed (Participants) | 20 | 18
  Week 2 | 147.4 [123.3 to 182.1] | 0.1 [0.1 to 0.1]
  Week 3 - Pre-Infusion | 113.6 [102.2 to 130.0] | 0.1 [0.1 to 0.1]
  Week 3 - Post-Infusion: number analyzed (Participants) | 19 | 0
  Week 3 - Post-Infusion | 1807.7 [1617.0 to 2105.5] |
  Week 4: number analyzed (Participants) | 19 | 19
  Week 4 | 361.9 [295.4 to 432.3] | 0.1 [0.1 to 0.1]
  Week 5: number analyzed (Participants) | 20 | 19
  Week 5 | 216.9 [174.6 to 254.2] | 0.1 [0.1 to 0.1]
  Week 6 - Pre-Infusion: number analyzed (Participants) | 19 | 19
  Week 6 - Pre-Infusion | 135.8 [112.2 to 164.5] | 0.1 [0.1 to 0.1]
  Week 6 - Post-Infusion: number analyzed (Participants) | 0 | 18
  Week 6 - Post-Infusion |  | 1643.5 [1483.3 to 2041.5]
  Week 7: number analyzed (Participants) | 18 | 19
  Week 7 | 95.9 [63.4 to 119.2] | 277.7 [240.7 to 318.2]
  Week 8: number analyzed (Participants) | 17 | 18
  Week 8 | 56.2 [35.5 to 82.7] | 158.0 [126.6 to 193.5]
  Week 9 - Pre-Infusion: number analyzed (Participants) | 19 | 19
  Week 9 - Pre-Infusion | 42.1 [21.1 to 56.8] | 98.7 [82.8 to 167.1]
  Week 9 - Post-Infusion: number analyzed (Participants) | 0 | 18
  Week 9 - Post-Infusion |  | 1717.8 [1446.9 to 2153.0]
  Week 10: number analyzed (Participants) | 17 | 19
  Week 10 | 37.8 [27.6 to 47.4] | 373.8 [302.3 to 416.0]
  Week 11: number analyzed (Participants) | 17 | 19
  Week 11 | 19.3 [10.4 to 28.1] | 217.2 [178.0 to 301.2]
  Week 12: number analyzed (Participants) | 19 | 19
  Week 12 | 13.4 [6.3 to 25.1] | 131.1 [106.3 to 215.3]
  Week 15: number analyzed (Participants) | 19 | 19
  Week 15 | 5.0 [1.9 to 10.9] | 42.1 [30.6 to 66.6]
  Week 18: number analyzed (Participants) | 19 | 19
  Week 18 | 2.1 [0.1 to 5.2] | 18.3 [9.0 to 45.6]
  Week 30: number analyzed (Participants) | 15 | 19
  Week 30 | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]

27. Secondary Outcome: Detectability of Antibody to VRC01 as Measured in Serum
Description: Assess the detectability of antibody to VRC01 in samples collected during study follow-up. Intended to be result from specimen at week 30 time point. Due to specimen availability, four participants in Arm A had results from specimens from the week 18 time point. Counts provided are number of participants with detectable anti-VRC01 antibody result.
Time Frame: Measured at week 30
Population: All participants with results for anti-VRC01 antibody. Two participants did not have results (one from each arm) due to being lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 19 | 19
Participants | 0 | 0

28. Secondary Outcome: Levels of T-cell Activation
Description: % CD4+ and CD8+ T-cells co-expressing human leukocyte antigen (HLA)-DR and CD38
  Not conducted as part of primary analysis and there are no future plans to assess this outcome. Samples were collected for this outcome in order to assess associations with virologic effects observed. Due to the lack of virologic effect observed, the study team has decided that this outcome is no longer of priority/interest and will be abandoned in favor of saving these samples for future research purposes.
Time Frame: Measured at screening, entry and weeks 1, 3, 4, 6, 7, 9, 10, 12, 15, 18 and 30
Population: Analysis not performed. See outcome measure description for reasoning.
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Levels of NK Cell Activation
Description: % NK cells expressing CD69 or CD95
  Not conducted as part of primary analysis and there are no future plans to assess this outcome. Samples were collected for this outcome in order to assess associations with virologic effects observed. Due to the lack of virologic effect observed, the study team has decided that this outcome is no longer of priority/interest and will be abandoned in favor of saving these samples for future research purposes.
Time Frame: Measured at screening, entry and weeks 1, 3, 4, 6, 7, 9, 10, 12, 15, 18 and 30
Population: Analysis not performed. See outcome measure description for reasoning.
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Plasma Levels of sCD163
Description: Not conducted as part of primary analysis and there are no future plans to assess this outcome. Samples were collected for this outcome in order to assess associations with virologic effects observed. Due to the lack of virologic effect observed, the study team has decided that this outcome is no longer of priority/interest and will be abandoned in favor of saving these samples for future research purposes.
Time Frame: Measured at screening, entry and weeks 1, 3, 4, 6, 7, 9, 10, 12, 15, 18 and 30
Population: Analysis not performed. See outcome measure description for reasoning.
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Plasma Levels of sCD14
Description: as for outcome 30
Time Frame: Measured at screening, entry and weeks 1, 3, 4, 6, 7, 9, 10, 12, 15, 18 and 30
Population: Analysis not performed. See outcome measure description for reasoning.
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Plasma Levels of Interleukin-6 (IL-6)
Description: as for outcome 30
Time Frame: Measured at screening, entry and weeks 1, 3, 4, 6, 7, 9, 10, 12, 15, 18 and 30
Population: Analysis not performed. See outcome measure description for reasoning.
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Plasma Levels of Human Soluble Tumor Necrosis Factor Alpha-receptor (sTNFαR)
Description: as for outcome 30
Time Frame: Measured at screening, entry and weeks 1, 3, 4, 6, 7, 9, 10, 12, 15, 18 and 30
Population: Analysis not performed. See outcome measure description for reasoning.
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Plasma Levels of Tumor Necrosis Factor Alpha (TNFα)
Description: as for outcome 30
Time Frame: Measured at screening, entry and weeks 1, 3, 4, 6, 7, 9, 10, 12, 15, 18 and 30
Population: Analysis not performed. See outcome measure description for reasoning.
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Plasma Levels of High-sensitivity C-reactive Protein (hsCRP)
Description: as for outcome 30
Time Frame: Measured at screening, entry and weeks 1, 3, 4, 6, 7, 9, 10, 12, 15, 18 and 30
Population: Analysis not performed. See outcome measure description for reasoning.
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: VRC01 Antibody Level Relative to Infusion Timing
Description: Summarize the pharmacokinetics (PK) of two infusions of VRC01 during study follow up - aligning the timing of PK samples/results to the respective VRC01 infusions for each Arm
Time Frame: Measured immediately after first infusion (and 1, 2, and 3 weeks after), and immediately after second infusion (and 1, 2, 3, 6 and 9 weeks after)
Population: Analysis of all participants with available results.
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
Number analyzed (Participants) | 20 | 20
ug/mL
  First dose - Post-Infusion: number analyzed (Participants) | 20 | 18
  First dose - Post-Infusion | 1726.2 [1492.5 to 1950.3] | 1643.5 [1483.3 to 2041.5]
  One week after first infusion: number analyzed (Participants) | 20 | 19
  One week after first infusion | 259.9 [213.0 to 297.5] | 277.7 [240.7 to 318.2]
  Two weeks after first infusion: number analyzed (Participants) | 20 | 18
  Two weeks after first infusion | 147.4 [123.3 to 182.1] | 158.0 [126.6 to 193.5]
  Three weeks after first infusion: number analyzed (Participants) | 20 | 19
  Three weeks after first infusion | 113.6 [102.2 to 130.0] | 98.7 [82.8 to 167.1]
  Second dose - Post-infusion: number analyzed (Participants) | 19 | 18
  Second dose - Post-infusion | 1807.7 [1617.0 to 2105.5] | 1717.8 [1446.9 to 2153.0]
  One week after second infusion: number analyzed (Participants) | 19 | 19
  One week after second infusion | 361.9 [295.4 to 432.3] | 373.8 [302.3 to 416.0]
  Two weeks after second infusion: number analyzed (Participants) | 20 | 19
  Two weeks after second infusion | 216.9 [174.6 to 254.2] | 217.2 [178.0 to 301.2]
  Three weeks after second infusion: number analyzed (Participants) | 19 | 19
  Three weeks after second infusion | 135.8 [112.2 to 164.5] | 131.1 [106.3 to 215.3]
  Six weeks after second infusion: number analyzed (Participants) | 19 | 19
  Six weeks after second infusion | 42.1 [21.1 to 56.8] | 42.1 [30.6 to 66.6]
  Nine weeks after second infusion: number analyzed (Participants) | 19 | 19
  Nine weeks after second infusion | 13.4 [6.3 to 25.1] | 18.3 [9.0 to 45.6]

ADVERSE EVENTS:
Time Frame: From first infusion through end of study follow up (the duration of the study is 30 weeks)
Description: The SAE Reporting Category, as defined in Version 2.0 of the DAIDS EAE Manual, was used for this study. At entry, signs, symptoms and laboratory values regardless of grade were reported. Post-entry, signs, symptoms and laboratory values grade ≥2, or those causing a change in treatment/ART, regardless of grade, were reported. Diagnoses identified on the study-specific list of diagnoses were recorded at entry and at all subsequent visits. Used DAIDS AE Grading Table, Version 2.0, November 2014
Arm/Group | Arm A: VRC01 Followed by Placebo | Arm B: Placebo Followed by VRC01
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 16/20 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: VRC01 Followed by Placebo (N=20) | Arm B: Placebo Followed by VRC01 (N=20)
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: VRC01 Followed by Placebo (N=20) | Arm B: Placebo Followed by VRC01 (N=20)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Eye movement disorder (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anogenital dysplasia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3
Reactive gastropathy (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 2
Fatigue (General disorders) | 1 | 2
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Acute sinusitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Alanine aminotransferase (Investigations) | 2 | 0
Aspartate aminotransferase (Investigations) | 1 | 1
Bilirubin conjugated abnormal (Investigations) | 2 | 0
Bilirubin conjugated increased (Investigations) | 1 | 1
Blood alkaline phosphatase abnormal (Investigations) | 1 | 0
Blood bilirubin abnormal (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 2
Blood creatinine abnormal (Investigations) | 2 | 3
Blood creatinine increased (Investigations) | 1 | 3
Blood glucose increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 1
Blood potassium increased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 6 | 10
Haemoglobin decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Burning sensation (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Psychogenic seizure (Psychiatric disorders) | 0 | 1
Genital lesion (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fixed drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No